CLINICAL TRIAL: NCT00001741
Title: Study of Vascular Responsiveness in Subjects With Polymorphisms of the Angiotensin II Type I Receptor Gene
Brief Title: Study of Inherited Changes of Receptors Located on Blood Vessels
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 980029; 98-H-0029
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-04

CONDITIONS: Cardiovascular Disease
Keywords: Angiotensin II Receptor; Polymorphism, Genetic; Vascular Tone; Angiotensin II; Losartan
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Losartan

INTERVENTIONS:
Drug: Losartan

SUMMARY:
The renin angiotensin system is a complex process involving hormones and enzymes that regulate blood volume and blood pressure. The hormone angiotensin II is responsible for making blood vessels narrow or constrict. Angiotensin II is found in the blood and can attach to special sites called receptors on blood vessel walls. These receptors are programmed to accept angiotensin II and cause a constriction of the blood vessel. This function is found in the genetic information of each individual person.

Occasionally patients have changes in their genes related to angiotensin II receptors. These changes may result in the receptors acting differently to angiotensin II, which may affect the function of blood vessels.

This study is designed to improve researchers understanding of the physiological effects on blood vessels associated with mutations of the genes responsible for angiotensin II receptor function.

DETAILED DESCRIPTION:
Polymorphisms in the genes encoding for various elements of the renin angiotensin system have been associated with cardiovascular disease. We have isolated novel alleles in the angiotensin II type I receptor gene. We propose this exploratory investigation to study the physiological effect of these mutations on vascular function in patients and family members who carry these rare alleles.

ELIGIBILITY:
Patients aged 21 or older with chronic orthostatic intolerance will be included.

There will be no exclusion from participation in the study on the basis of ethnicity/race.

Patients will be recruited in the Cardiology Branch outpatient clinic, Dr. David Goldstein (Chief Neurocardiology Section, NINDS, NIH), or from outside physicians.

Children will be excluded from the study because of inability in obtaining informed consent.

Cognitively impaired individuals, prisoners, or other institutionalized persons will not be able to participate.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 1997-11; Study Completion 2003-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Rigat B, Hubert C, Alhenc-Gelas F, Cambien F, Corvol P, Soubrier F. An insertion/deletion polymorphism in the angiotensin I-converting enzyme gene accounting for half the variance of serum enzyme levels. J Clin Invest. 1990 Oct;86(4):1343-6. doi: 10.1172/JCI114844. PMID 1976655
- [Background] Cambien F, Poirier O, Lecerf L, Evans A, Cambou JP, Arveiler D, Luc G, Bard JM, Bara L, Ricard S, et al. Deletion polymorphism in the gene for angiotensin-converting enzyme is a potent risk factor for myocardial infarction. Nature. 1992 Oct 15;359(6396):641-4. doi: 10.1038/359641a0. PMID 1328889
- [Background] Alderman MH, Madhavan S, Ooi WL, Cohen H, Sealey JE, Laragh JH. Association of the renin-sodium profile with the risk of myocardial infarction in patients with hypertension. N Engl J Med. 1991 Apr 18;324(16):1098-104. doi: 10.1056/NEJM199104183241605. PMID 1759997